CLINICAL TRIAL: NCT03628677
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of AB154 Monotherapy and Combination Therapy in Participants With Advanced Malignancies
Brief Title: A Study to Evaluate the Safety and Tolerability of AB154 in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB154CSP0001
Record Dates: First submitted 2018-07-26; First posted 2018-08-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Unspecified, Adult
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Intervention Model Description: Dose Escalation Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Domvanalimab Monotherapy (Experimental): Varying Doses of domvanalimab Monotherapy
  Interventions: Drug: Domvanalimab
- Domvanalimab + zimberelimab Q2W Combination Therapy (Experimental): Varying Doses of domvanalimab in Combination With Varying Doses of zimberelimab
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Domvanalimab + zimberelimab Q3W Combination Therapy (Experimental): Varying Doses of domvanalimab in Combination With Varying Doses of zimberelimab
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Domvanalimab + zimberelimab Q4W Combination Therapy (Experimental): Varying Doses of domvanalimab in Combination With Varying Doses of zimberelimab
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Domvanalimab and Zimberelimab Q6W combination therapy (Experimental): Varying Doses of domvanalimab in Combination With Varying Doses of zimberelimab
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Fixed dose Domvanalimab Q3W or Q4W and Zimberelimab Q3W, Q4W (Experimental): Varying Doses of domvanalimab in Combination With Varying Doses of zimberelimab
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab

INTERVENTIONS:
Drug: Domvanalimab — Domvanalimabis a fully human immunoglobulin G1 (IgG1) monoclonal antibody targeting human TIGIT
  Other Names: AB154
Drug: Zimberelimab — Zimbererlimab is a fully human immunoglobulin G4 (IgG4) monoclonal antibody targeting human PD-1
  Other Names: AB122
  Arms: Domvanalimab + zimberelimab Q2W Combination Therapy; Domvanalimab + zimberelimab Q3W Combination Therapy; Domvanalimab + zimberelimab Q4W Combination Therapy; Domvanalimab and Zimberelimab Q6W combination therapy; Fixed dose Domvanalimab Q3W or Q4W and Zimberelimab Q3W, Q4W

SUMMARY:
This is a Phase 1, multicenter, open-label, dose-escalation study to evaluate the safety, tolerability, PK, PD, and clinical activity of domvanalimab (AB154) as monotherapy and in combination with zimberelimab (AB122) in participants with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Male or female participants ≥ 18 years of age at the time of screening
* Negative serum pregnancy test at screening and prior to dosing on Cycle 1 Day 1; negative serum or urine pregnancy test on the first day of each subsequent treatment period
* Participants with any pathologically confirmed solid tumor type for which no standard of care therapy exists
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The measurable lesion must be outside of a radiation field if the participant received prior radiation
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 7. Confirmation that an archival tissue sample is available and ≤ 6 months old; if not, a new biopsy of a tumor must be obtained 8. Immunosuppressive doses of systemic medications, such as corticosteroids or absorbed topical corticosteroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks (14 days) before investigational product administration. Physiologic doses of corticosteroids ≤ 10 mg/day of prednisone or its equivalent may be permitted
* Prior surgery that required general anesthesia or other major surgery as defined by the Investigator must be completed at least 4 weeks before investigational product administration
* Negative tests for hepatitis B surface antigen, hepatitis C virus antibody (or hepatitis C qualitative ribonucleic acid [RNA; qualitative]), and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Adequate organ and marrow function

Exclusion Criteria:

* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of investigational product
* Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of investigational product hazardous (eg, interstitial lung disease, active infections requiring antibiotics, recent hospitalization with unresolved symptoms)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of domvanalimab as monotherapy and in combination with zimberelimab.
* Participants who require a Legally Authorized Representative (LAR) to provide informed consent on their behalf.
* Any active autoimmune disease or a documented history of autoimmune disease or history of a syndrome that required systemic steroids or immunosuppressive medications, except for vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study
* Prior malignancy active within the previous year except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer
* Has had prior chemotherapy, targeted small-molecule therapy, immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer), biologic agents or radiation therapy within 4 weeks (or 5 half-lives) prior to Day 1 or has not recovered from AEs due to a previously administered agent
* Use of other investigational drugs within 28 days or at least 5 half-lives before investigational product administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | From First Dose Date to 100 Days After Last Dose
  Number of Participants Treated with domvanalimab or domvanalimab in Combination with zimberelimab with Treatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
AB154 Peak Plasma Concentration (Cmax) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Peak Plasma Concentration (Cmax) of domvanalimab
Zimberelimab Peak Plasma Concentration (Cmax) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Peak Plasma Concentration (Cmax) of zimberelimab
Domvanalimab Time of Peak Concentration (Tmax) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Time of Peak Concentration (Tmax) of domvanalimab
Zimberelimab Time of Peak Concentration (Tmax) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Time of Peak Concentration (Tmax) of zimberelimab
Domvanalimab Area Under the Plasma Concentration Versus Time Curve (AUC) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Area Under the Plasma Concentration Versus Time Curve (AUC) of domvanalimab
Zimberelimab Area Under the Plasma Concentration Versus Time Curve (AUC) | Day 1 (sequential), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29 (sequential), Day 30, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 113, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Area Under the Plasma Concentration Versus Time Curve (AUC) of zimberelimab
Immunogenicity Indicators: Anti-Drug Antibodies (ADA) | Day 1, Day 15, Day 29, Day 43, Day 57, Day 85 and 30 Days After Last Dose, up to 52 weeks
  Number of Participants who Develop Antidrug Antibodies to AB154 and/or AB122
Overall Response Rate | First Dose Date to Progression or Last Tumor Assessment, up to 1 year
  Number of Participants with Complete or Partial Response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.1
Duration of Response | Start Date of Response to First Progression/Death, up to 1 year
  Time at Which Response Criteria are Met for Complete Response or Partial Response (Whichever Occurs First) Until the First Date of Recurrence, Progression or Death per RECIST v1.1
Disease Control Rate | First Dose Date to First Progression/Death, up to 1 year
  Number of Participants with Complete Response, Partial Response, or Stable Disease for Greater Than 6 Months per RECIST v1.1
Progression Free Survival | First Dose Date to First Progression/Death, up to 1 year
  Number of Participants Without Disease Progression per RECIST v1.1
Overall Survival | First Dose Date to Date of Death, up to 1 year
  Overall Survival Rate, Defined as Time Between First Dose Date and Date of Death

OTHER OUTCOMES:
Domvanalimab Receptor Occupancy | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Receptor Occupancy May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Domvanalimab Immunophenotyping | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Immunophenotyping May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Domvanalimab Gene Expression | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Gene Expression May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Domvanalimab Cytokines | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Cytokines May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples.
.Zimberelimab Receptor Occupancy | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Receptor Occupancy May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Zimberelimab Immunophenotyping | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Immunophenotyping May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Zimberelimab Cytokines | : Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141 and 30 Days After Last Dose, up to 52 weeks
  Cytokines May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples
Zimberelimab Gene Expression | Day 1, Day 3, Day 8, Day 15, Day 22, Day 29, Day 31, Day 36, Day 43, Day 57, Day 64, Day 85, Day 106, Day 141, and 30 Days After Last Dose, up to 52 weeks
  Gene Expression May be Summarized by Dose Group and Subject Over Time by Aggregating Data From Exploratory Biomarkers Collected From Peripheral Blood Samples

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (10):
- United States (6):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Affinity Health-Hope and Healing Cancer Services, LLC, Hinsdale, Illinois
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - START, San Antonio, Texas
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane, Washington
- Australia (4):
  - The Kinghorn Cancer Centre - St Vincent Public Hospital, Darlinghurst, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Icon Cancer Care Brisbane, South Brisbane, Queensland
  - Olivia Newton-John Cancer Research Institute-Austin Hostipal, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents [e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)] upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: AB154CSP0001 - Public Website — https://trials.arcusbio.com/study/?id=AB154CSP0001